CLINICAL TRIAL: NCT03662854
Title: Phase 1, Randomized, Double-Blind, Vehicle-Controlled Study of Safety and Tolerability of Hair Stimulating Complex (HSC) in Female Subjects With Female Pattern Hair Loss
Brief Title: Safety and Tolerability of Hair Stimulating Complex (HSC) in Female Pattern Hair Loss
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Histogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-HIS002-US
Record Dates: First submitted 2018-08-14; First posted 2018-09-10 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2018-08

CONDITIONS: Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: Placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinding
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hair Stimulating Complex (Experimental): Hair Stimulating Complex (HSC) is derivative of hypoxia-induced multipotent cell conditioned media enriched for certain key growth factors
  Interventions: Biological: Hair Stimulating Complex (HSC)
- Phosphate Buffered Saline (Placebo Comparator): Phosphate Buffered Saline
  Interventions: Other: Phosphate Buffered Saline

INTERVENTIONS:
Biological: Hair Stimulating Complex (HSC) — Patients will receive 2 mL of HSC separated by 6 weeks (total of 4 mL of HSC)
  Arms: Hair Stimulating Complex
Other: Phosphate Buffered Saline — Patients will receive 2 mL of Phosphate Buffered Saline separated by 6 weeks (total of 4 mL of Phosphate Buffered Saline)
  Arms: Phosphate Buffered Saline

SUMMARY:
This double-blind placebo-controlled study will assess the tolerability, feasibility, and pharmacodynamics of intradermal Hair Stimulating Complex (HSC) in up to 18 of 27 women with Ludwig 1 or 2 classification or the Savin Frontal classification of hair loss. Safety measures include vital signs, dermatological examination of the scalp, pre- and post-dose blood and urine collection, as well as Investigator Global Assessments and subject self assessments throughout the 22-week study.

DETAILED DESCRIPTION:
The study is a double-blind, placebo-controlled, randomized single site trial. The study is to be conducted in La Jolla, CA and is primarily designed to evaluate safety in the clinical application of injected HSC by assessing the tolerability of HSC, as well as the volume that can be delivered safely in the intradermal region of the scalp using a syringe with 31-gauge 1.75 mm length needle. The main study (18 weeks) involves the two treatment time points, collection of lab samples (blood/urine) for screening, and before and after the two treatment time points. Six of the seven total visits (including screening) in the study are conducted in the first 18 weeks. The final visit is for investigator monitoring, global photographs and final lab collection 30 days after the 18-week evaluation point. A 2 year follow up questionnaire will be sent to the patient to collect additional safety information. Additional dermatological exam of the scalp, as well as Subject and Investigator Assessments will also be assessed. The secondary goal of the study will be to explore whether an efficacy signal of the change in hair growth can be detected using an independent panel of physician's comparing global photographs taken at baseline to week 18 (and baseline to week 22), for changes.

ELIGIBILITY:
Inclusion Criteria:

* Female, 40-70 years of age.
* A healthy scalp with no cutaneous disorder.
* Good general health.
* Must fulfill the Ludwig I or II classification or Savin classification of frontal hair loss (see Appendix 1).
* Willing and able to comply with scheduled visits (6 visits in 22 weeks).
* Willing to maintain the same hair style and color during the study period.
* Subjects not already using any over-the-counter or prescription hair/scalp treatments, must be willing to refrain from starting use of any new hair/scalp products other than the provided study product for the duration of the study.
* Willingness to have blood and urine samples taken before and after each of the two treatments to evaluate overall systemic effect and also at Weeks 18 and 22. Also willing to give additional serum samples at each collection for long-term storage and immunogenicity testing by Histogen to components in HSC.
* Be able to speak and read English to the standard required to provide written informed consent and to cooperate with the study staff.
* Female subjects will be either of non-childbearing potential defined as:

  1. Having no uterus
  2. No menses for at least 12 months. Or; (WOCBP) women of childbearing potential must agree to use an effective method of birth control during the course of the study, such as:

  <!-- -->

  1. Oral contraceptive pill, injection, implant, patch, vaginal ring, intrauterine device
  2. Intrauterine coil
  3. Bilateral tubal ligation
  4. Barrier method used with an additional form of contraception (e.g., sponge, spermicide or condom)
  5. Abstinence (If practicing abstinence must agree to use barrier method described above (4) if becomes sexually active).
  6. Vasectomized partner (Must agree to use barrier method described above (4) if becomes sexually active with non-vasectomized).

     -

     Exclusion Criteria:
* Known sensitivity to any of the test material ingredients.
* History of keloid formation or hyperpigmentation.
* Pregnant, planning pregnancy or breastfeeding during the course of the study.
* A history of any acute or chronic illness that in the opinion of the investigators might confound the results of the study including some drugs or medications.
* Active skin diseases (e.g. Eczema, seborrheic dermatitis, psoriasis, skin cancer, sun damaged skin with actinic keratosis on scalp, excessive number and size of seborrheic keratosis, etc.).
* Routine high dosage use of anti-inflammatory medications (aspirin, ibuprofen, corticosteroids), immunosuppressive drugs or antihistamine medications (Note that steroid nasal spray / drops and/or topical steroids administered to the eye(s) are not exclusion criteria, and that a daily dose of 81 - 325mg aspirin is also permitted).
* (Auto-) Immunological disorders such as HIV positive, alopecia areata, and systemic lupus erythematosus.
* Participation in any clinical study within one month prior to enrollment or planned participation in any clinical trial during the duration of their participation in this study.
* Treatment with an experimental or investigative drug or product within the last 3 months.
* Moderate/severe Seborrheic dermatitis (scalp).
* Damaged skin in or around test sites (including sunburn, uneven skin tones, tattoos, scars or other disfiguration of the test site).
* Use of any over-the-counter or prescription hair/scalp treatments for less than 6 months from date subject would start study, including finasteride or minoxidil.
* Discontinuation of the use of an over-the-counter or prescription hair/scalp treatments within the last 6 months
* Use of laser or light device for the scalp for purposes of hair growth within the last 6 months or any plans to use these devices during the duration of the study.
* History of hair transplantation surgery during the last 6 months.
* Currently using hair system or wig and/or unwilling to refrain from use throughout the duration of the study.
* History of malignancy, other than non-melanoma skin cancer. Any condition for which the Investigator determines that the subject could be placed under undue hazard.
* Known allergy to rice.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2021-01-21 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events due to HSC | Continuous for 22 weeks after first dose
  Safety and tolerability of HSC by comparing adverse events to baseline

SECONDARY OUTCOMES:
Investigator Assessments of Global Photographs compared to baseline | Day 1, Week 18 and 22
  Investigator Assessments of Global Photographs compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Cosmetic Laser Dermatology, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No